CLINICAL TRIAL: NCT02139670
Title: Thrombin Generation and Gestational Outcome in Women With Recurrent Pregnancy Loss
Brief Title: Thrombin Generation and Gestational Outcome
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elias mazen, Director of Internal medicine, HaEmek Medical Center, Israel
Other Study IDs: thrombin generation- pregnancy
Record Dates: First submitted 2013-08-26; First posted 2014-05-15 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Thrombophilia
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — 4 cc of serum will be retain until all blood samples will be collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pregnant womens

SUMMARY:
In total 120 pregnant women's with history of recurrent miscarriages, are planned for inclusion in this trial. After signing an informed consent a blood sample will be obtained from each participant. The investigators will measure the thrombin generation in plasma assessed by the calibrated automated thrombogram (CAT). The relation between pregnancy outcome and thrombin measurements will be determined

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* signed inform consent
* first trimester
* two early miscarriages(before week 10) or one later abortions (after week 10)

Exclusion Criteria:

* Chronic treatment with aspirin or other anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women with recurrent miscarriages undergoing investigation for Thrombophilia .
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
pregnancy outcome | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: mazen elias, prof, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Haemek medical center, Afula, Israel